CLINICAL TRIAL: NCT06230458
Title: Care Evaluation Study of the Fractional Exhaled Nitric Oxide (FeNO)- Test as add-on Test in the Diagnostic Work-up of Asthma
Brief Title: Fractional Exhaled Nitric Oxide (FeNO)- Test as add-on Test in the Diagnostic Work-up of Asthma
Acronym: INFERNO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Franciscus Gasthuis & Vlietland (Hospital) (Other)
Collaborators: OLVG (Network)
Responsible Party: Principal Investigator, Hanna Kuiper- van der Valk, Principal investgator, Franciscus Gasthuis & Vlietland (Hospital)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: R23.005
Record Dates: First submitted 2023-12-13; First posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Diagnosis; Asthma
Keywords: Asthma; Diagnostics; FeNO; Bronchial provocation test; Burdesome; cost-effectiveness
MeSH Terms: conditions — Disease; Asthma | interventions — Fractional Exhaled Nitric Oxide Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Asthma patients without reversibility (Other): Asthma patients without reversibility
  Interventions: Diagnostic Test: FeNO-test

INTERVENTIONS:
Diagnostic Test: FeNO-test — Fractional Exhaled Nitric Oxide (FeNO)- test

SUMMARY:
The Global Initiative of Asthma Guideline (GINA) recommends a flowchart to diagnose asthma with first-step spirometry with reversibility and a bronchial challenge test (BPT) with histamine or methacholine as a second step.

This multi-center prospective care evaluation study compares the 'standard asthma diagnostic work-up' (spirometry with reversibility and BPT) to the 'new asthma diagnostics work-up' (FeNO-test as an intermediate step between the spirometry with reversibility and the BPT), intending to determine the impact of the FeNO-based strategy, in terms of the number of avoided BPTs, cost-effectiveness and reduced burden to the patient and health care.

The cost reduction of incorporating the FeNO-test in the new diagnostic algorithm will be established by the number of theoretically avoided BPT. The decrease in burden will be studied by calculating differences in the Visual Analogue Scale (VAS) -score and Asthma Quality of Life Questionnaire (AQLQ) -score after the BPT and FeNO-test with an independent T-test. The accuracy of the FeNO-test will be calculated by comparing the FeNO-test outcomes to the (gold standard) BPTs outcomes in terms of sensitivity and specificity.

DETAILED DESCRIPTION:
Background Asthma is a common disease characterized by chronic inflammation of the lower airways, bronchial hyperactivity, and (reversible) airway obstruction. The Global Initiative of Asthma Guideline (GINA) recommends a flowchart to diagnose asthma with first-step spirometry with reversibility and a bronchial challenge test (BPT) with histamine or methacholine as a second step. The BPT is considered burdensome, time-consuming for patients and staff, can cause side effects, and is expensive. In addition, this test strongly encumbers lung function capacity. Elevated Nitric Oxide (NO) is associated with airway eosinophilic inflammation in asthma patients and can be measured in exhaled air with the Fractional exhaled (Fe) NO-test. This low-burden FeNO-test could be used as an 'add-on' test in asthma diagnostics.

Methods/analysis This multi-center prospective care evaluation study compares the 'standard asthma diagnostic work-up' (spirometry with reversibility and BPT) to the 'new asthma diagnostics work-up' (FeNO-test as an intermediate step between the spirometry with reversibility and the BPT), intending to determine the impact of the FeNO-based strategy, in terms of the number of avoided BPTs, cost-effectiveness and reduced burden to the patient and health care. The accuracy of the FeNO-test is included for verification.

The cost reduction of incorporating the FeNO-test in the new diagnostic algorithm will be established by the number of theoretically avoided BPT. The decrease in burden will be studied by calculating differences in the Visual Analogue Scale (VAS) -score and Asthma Quality of Life Questionnaire (AQLQ) -score after the BPT and FeNO-test with an independent T-test. The accuracy of the FeNO-test will be calculated by comparing the FeNO-test outcomes to the (gold standard) BPTs outcomes in terms of sensitivity and specificity.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old visiting the outpatient clinic pulmonology with the suspicion of asthma will be asked to participate in this study. For reasons of external validity and generalizability of the study results, it was decided not to exclude subgroups such as smokers or obese patients.

Exclusion Criteria:

* Patients with already diagnosed asthma are not allowed to participate.
* The inclusion of patients with respiratory infections <3 weeks ago will be postponed to >3 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Number of provocation tests per year | 1 year

SECONDARY OUTCOMES:
Costs per year | 1 year
Burden for the patient per through study completion | 1 year
Accurancy FeNO-test through study completion | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Hanna Kuiper-van der Valk, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No
It is not yet known if there will be a plan to make IPD available.